CLINICAL TRIAL: NCT05263362
Title: An Integrated Optimization of Surgery and Radiotherapy Techniques to Improve Cosmetic Outcome and Quality of Life in Breast Conserving Therapy for Breast Cancer Patients.
Brief Title: An Integrated Optimization of Surgery and Radiotherapy Techniques to Improve Cosmetic Outcome and Quality of Life in Breast Conserving Therapy for Breast Cancer Patients (STARLINGS Study)
Acronym: STARLINGS
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Albert Schweitzer Ziekenhuis, Netherlands (Other)
Responsible Party: Principal Investigator, E. (Euphemia) A.M. Froklage, MD, PhD, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2021-0829
Record Dates: First submitted 2022-01-12; First posted 2022-03-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Fibrosis; Breast Cancer; Breast Cancer Female; Breast Neoplasms; Breast Carcinoma in Situ; Breast Carcinoma
Keywords: Fibrosis; Cosmetic outcome; Quality of life; Oncoplastic breast surgery; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STARLINGS study population: The study population consists of breast cancer patients who were treated with breast conserving therapy (BCT) at one of the four participating hospitals (Erasmus MC, Albert Schweitzer hospital, Maasstad hospital and Franciscus hospital Gasthuis and Vlietland), for non-metastatic, histological proven invasive breast cancer or DCIS between 2016 and 2020 (at time of inclusion in 2022 respectively 6 to 2 years after treatment), and subsequently received adjuvant (whole breast) irradiation (WBI), with or without boost, at the Erasmus MC as part of their BCT.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — At one timepoint patients will get physical examination of the breasts, medical photographs will be taken, and they will fill in five questionnaires about satisfaction of the breasts, quality of life and general health.

SUMMARY:
To assess the role of different combinations of (oncoplastic) surgery and radiotherapy techniques as risk factors for moderate to severe fibrosis and for moderate to poor cosmetic outcome.

DETAILED DESCRIPTION:
The primary objectives of this study are to assess the role of different combinations of (oncoplastic) surgery and radiotherapy techniques as risk factors for moderate to severe fibrosis and for moderate to poor cosmetic outcome. Based on these insights predictive models for the development of moderate to severe fibrosis and moderate to poor cosmetic outcome will be developed. Second, the relation between the presence and severity of fibrosis, cosmetic outcome and different QoL domains and symptoms will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years
* History of BCT with adjuvant radiation therapy for non-metastatic, histologically proven invasive breast cancer or DCIS. In light of BCT adjuvant systemic treatment (i.e. endocrine therapy, chemotherapy and immune therapy) is allowed.
* Operated between 1st of January 2016 and 31th of December 2020
* Treated according to the currently applied dose fractionation schedules, i.e. whole breast radiotherapy (22, 23), with or without boost
* Adequate understanding of the Dutch language and written informed consent

Exclusion Criteria:

* Any breast surgery or re-irradiation on the breast area after BCT
* Progression of disease (and additional treatment) since BCT
* Patients who received partial breast irradiation
* Current pregnancy or breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of breast cancer patients who were treated with breast conserving therapy (BCT) at one of the four participating hospitals (Erasmus MC, Albert Schweitzer hospital, Maasstad hospital and Franciscus hospital Gasthuis and Vlietland), for non-metastatic, histological proven invasive breast cancer or DCIS between 2016 and 2020 (at time of inclusion in 2022 respectively 6 to 2 years after treatment), and subsequently received adjuvant radiotherapy of the whole breast at the Erasmus MC as part of their BCT.
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Fibrosis of the breast as measured by CTCAE v5 scale | 2-6 years after breast conserving treatment. 1 point of measurement.
  Fibrosis will be graded by the researcher using the CTCAE v5 scale.
  On the CTCAE scale of superficial soft tissue fibrosis:
  Grade 0 = no fibrosis, Grade 1 = mild induration, able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up), Grade 2 = Moderate induration, able to slide skin, unable to pinch skin; limiting instrumental ADL, Grade 3 = Severe induration; unable to slide or pinch skin; limiting joint or orifice movement (e.g., mouth, anus); limiting self care ADL, Grade 4 = Generalized; associated with signs or symptoms of impaired breathing or feeding, Grade 5 = Death.
  We are planning to score fibrosis of the breast as none/mild (grade 0-1) or moderate/severe (grade 2-3).
Cosmetic outcome as measured by 9-item questionnaire | 2-6 years after breast conserving treatment. 1 point of measurement.
  Cosmetic outcome will be evaluated by means of a 9-item cosmetic patient questionnaire filled out by the patient with scoring on a four point scale (range from 'excellent' to 'poor' per item).
Cosmetic outcome as measured by BCCT.core software | 2-6 years after breast conserving treatment. 1 point of measurement.
  Patients' photographs of the breasts will be taken. With the use of BCCT.core software from The Breast Research group (INESC TEC, the Faculdade de Medicina da Universidade do Porto) cosmetic outcome will be assessed.

SECONDARY OUTCOMES:
Quality of life, as measured by BREAST-Q | 2-6 years after breast conserving treatment. 1 point of measurement.
  Which includes the following domains: psychosocial well being, sexual well being, satisfaction with the breasts, physical well being, adverse effects of radiation.
  All domains are scored 0 to 100 points, higher points means a better outcome.
Quality of life, as measured by EORTC Quality of Life Questionnaires-C30 | 2-6 years after breast conserving treatment. 1 point of measurement.
  Which include functional domains, global health status and symptom scales.
  For functional domains and global health status, scores range from 0 to 100. Higher scores means a better level of functioning. For symptoms scales, scores range from 0 to 100. Higher scores represent a greater degree of symptoms.
Quality of life, as measured by EORTC Quality of Life Questionnaires-B23 | 2-6 years after breast conserving treatment. 1 point of measurement.
  Which include functional domains, global health status and symptom scales.
  For functional domains and global health status, scores range from 0 to 100. Higher scores means a better level of functioning. For symptoms scales, scores range from 0 to 100. Higher scores represent a greater degree of symptoms.
Quality of life, as measured by EQ-5D-5L - five dimensions | 2-6 years after breast conserving treatment. 1 point of measurement.
  The EQ-5D-5L include five questions about five dimensions: mobility, self-care, daily activities, pain/discomfort and anxiety/depression.
  For each dimension, participants choose one of five levels that best fits their health on that day (from 'no problem'= 1 to 'unable/extreme'= 5). The numbers chosen for the five dimensions are combined to give a 5 digit score (minimum score = 11111 maximum score = 55555).
Quality of life, as measured by EQ-5D-5L - VAS | 2-6 years after breast conserving treatment. 1 point of measurement.
  The EQ-5D-5L include, apart from the five questions about five dimensions (see above), a visual analogue scale (VAS).
  The VAS provides rating of the participant's health on a scale from 0 ('the worst health you can imagine') to 100 ('the best health you can imagine').

CONTACTS AND LOCATIONS:
Overall Officials: R.A. Nout, Professor, Study Director — Erasmus Medical Center; E.A.M. Froklage, MD, PhD, Principal Investigator — Erasmus Medical Center; M.B.E. Menke-Pluijmers, MD, PhD, Principal Investigator — Albert Schweitzer Hospital
Locations (4):
- Netherlands (4):
  - Albert Schweitzer hospital, Dordrecht
  - Erasmus Medical Center, Rotterdam
  - Maasstad hospital, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Notenboom MCAW, Klem TMAL, Contant CME, Ribbe SP, Franckena M, Penninkhof JJ, Koppert LB, Plaisier PW, Mureau MAM, van Werkhoven ED, van der Veen FJC, de Kraker M, Nout RA, Menke-Pluijmers MBE, Froklage FE. The association between breast fibrosis, cosmetic outcomes, and long-term health-related quality of life after breast-conserving therapy: a multicenter cross-sectional observational cohort study. Breast. 2025 Oct;83:104541. doi: 10.1016/j.breast.2025.104541. Epub 2025 Jul 14. PMID 40774221